CLINICAL TRIAL: NCT00869570
Title: Neoadjuvant Radiotherapy Combined With Capecitabine and Sorafenib in Patients With Advanced, K-ras Mutated Rectal Cancer. A Multicenter Phase I/IIa Trial.
Brief Title: External-Beam Radiation Therapy, Capecitabine, and Sorafenib in Treating Patients With Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 41/08; SWS-SAKK-41-08; 2008-006312-38 (EudraCT Number); CDR0000634955 (Other: www.clinicalcollections.org)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Sorafenib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A: Sorafenib & Capecitabine & RT (Experimental): Sorafenib: day 1 to 33 (5 weeks, including Saturday and Sunday) every 24 hours, immediately or within two hours after RT according to the dose escalation table during phase I, and the recommended dose during phase IIa. The intake stops at the last day of RT. On nonradiotherapy days (e.g. Saturday, Sunday), the tablets have to be taken at the same time as during the week.
  * Capecitabine: day 1 to 33 (5 weeks, including Saturday and Sunday) according to dose escalation table during phase I, and at the recommended dose during phase IIa. The intake stops in the evening of the last day of RT.
  * External beam RT: Monday through Friday for 5 weeks starting on day 1 (daily fraction 1.8 Gy, final dose 45 Gy) each day at the same time (e.g. 11:00 a.m. daily).
  * Surgery: 6 weeks (± 1 week) after radiochemotherapy (RCT) has been completed
  Interventions: Drug: capecitabine; Drug: sorafenib tosylate; Radiation: radiation therapy

INTERVENTIONS:
Drug: capecitabine — Phase II: 2 x 825 mg/m2 per day (during 5 weeks)
  Other Names: XELODA
Drug: sorafenib tosylate — Phase II: 1 x 400 mg per day (during 5 weeks)
  Other Names: BAY 43-9006
Radiation: radiation therapy — Phase II: 1.8 Gy per day in 25 fractions (during 5 weeks)

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving radiation therapy together with capecitabine and sorafenib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I/II trial is studying the side effects and best dose of capecitabine when given together with sorafenib and external-beam radiation therapy and to see how well it works in treating patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recommended dose of neoadjuvant capecitabine when given together with sorafenib tosylate and external-beam radiotherapy in patients with K-ras mutated, locally advanced rectal cancer. (Phase I)
* Assess the efficacy and safety of this regimen in these patients. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of capecitabine followed by a phase II study.

Patients receive oral capecitabine twice daily and oral sorafenib tosylate once daily on days 1-33. Patients also undergo external-beam radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33. Approximately 6 weeks after completion of neoadjuvant therapy, patients undergo surgery.

After completion of study therapy, patients are followed at 8 weeks and then periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally advanced adenocarcinoma of the rectum (with or without nodal involvement) requiring surgery

  * Stage mrT3-4, and/or mrN1-2, M0 disease
* Tumor with K-ras gene mutation as assessed locally
* No distant metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL
* Creatinine clearance ≥ 50mL/min
* AST ≤ 2.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* PT/INR or PTT ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 12 months after completion of study therapy
* Is compliant and geographic proximity allows for proper staging and follow-up
* No other malignancy within the past 5 years except adequately treated cervical carcinoma in situ or localized nonmelanoma skin cancer
* No psychiatric disorder that would preclude understanding study-related information, giving informed consent, or complying with oral drug intake
* No clinically significant (i.e., active) cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease, or cardiac arrhythmia [even if controlled with medication]) or myocardial infarction within the past 12 months
* No uncontrolled hypertension
* No evidence or history of bleeding diathesis
* No lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* No serious or underlying condition (e.g., active autoimmune disease, uncontrolled diabetes, or uncontrolled infection) that, in the judgement of the investigator, could preclude the ability of the patient to participate in the study
* No known hypersensitivity to study drugs or to any other component of the study drugs

PRIOR CONCURRENT THERAPY:

* No prior treatment for rectal cancer
* No prior organ allografts
* More than 4 weeks since prior major surgery other than colostomy
* More than 30 days since prior treatment in a clinical trial
* No other concurrent experimental drugs or anticancer therapy
* No concurrent brivudine, lamivudine, ribavirin, or any other nucleoside analogue
* No concurrent drugs contraindicated for use with the study drugs
* No other concurrent radiotherapy
* No concurrent anticoagulation therapy other than low molecular weight heparin

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-03; Primary Completion 2013-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity of the treatment combination (Phase I) | during trial treatment (12 weeks)
Pathological near complete or complete tumor response (Dworak grade 3 and 4) (Phase II) | after trial treatment (approx. 12 weeks).

SECONDARY OUTCOMES:
R0 and R1 resection | after trial treatment (approx. 12 weeks)
Postoperative complications | within 8 weeks after surgery
Time to distant failure | during 3 years follow-up.
Disease-free survival | during 3 years follow-up.
Adverse events as assessed by NCI CTCAE v3.0 | during trial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Roger von Moos, MD, Study Chair — Kantonsspital Graubuenden
Locations (18):
- Szent Laszlo Korhaz, Budapest, Hungary
- Switzerland (17):
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital, Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneva HUG, Geneva
  - Kantonsspital Luzern, Lucerne
  - OnkoZentrum Luzern at Klinik St. Anna, Lucerne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum - Klinik im Park, Zurich
  - Stadtspital Triemli, Zurich
  - Onkozentrum Hirslanden, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] von Moos R, Koeberle D, Schacher S, Hayoz S, Winterhalder RC, Roth A, Bodoky G, Samaras P, Berger MD, Rauch D, Saletti P, Plasswilm L, Zwahlen D, Meier UR, Yan P, Izzo P, Klingbiel D, Bartschi D, Zaugg K; Swiss Group for Clinical Cancer Research (SAKK). Neoadjuvant radiotherapy combined with capecitabine and sorafenib in patients with advanced KRAS-mutated rectal cancer: A phase I/II trial (SAKK 41/08). Eur J Cancer. 2018 Jan;89:82-89. doi: 10.1016/j.ejca.2017.11.005. Epub 2017 Dec 11. PMID 29241084